CLINICAL TRIAL: NCT04294511
Title: A Phase Ⅱ ,Open-label ,Single Institution Study to Investigate the Efficacy and Safety of Camrelizumab in Combination With Neoadjuvant Chemotherapy in the Treatment of Locally , Resectable Osteosarcoma
Brief Title: Study of Camrelizumab in Combination With Neoadjuvant Chemotherapy in the Treatment of Osteosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jin Wang,MD, Director of bone and soft tissue, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-STS-II-002
Record Dates: First submitted 2020-02-26; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — camrelizumab; Neoadjuvant Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): camrelizumab in combination with adriamycin, cisplatin, ifosfamide and methotrexate
  Interventions: Drug: Camrelizumab in Combination With Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Camrelizumab in Combination With Neoadjuvant Chemotherapy — camrelizumab in combination with adriamycin, cisplatin, ifosfamide and methotrexate
  Other Names: PD-1 inhibitor

SUMMARY:
This study is a open-lable, , single center, phase II clinical study. Target population is patients with locally resectable osteosarcoma. Study objective is to compare the efficacy and safety of camrelizumab in combination with adriamycin, cisplatin, ifosfamide and methotrexate in study population in China. Camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
In this study, eligible subject will be enrolled into study arm to accept study treatment. Treatment cycles of chemotherapy will be at most 9 cycles which will be decided by investigators. The percentage of the patient with tumor cell necrosis rate >90% determined by the Independent Review Committee (IRC) will be the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14 to 65 year old
2. Eastern Cooperative Oncology Group performance status 0-1
3. Histopathologically diagnosed osteosarcomas (except for paraspesarcomas ), have been evaluated in patients have achieved normative resection with neoadjuvant chemotherapy
4. Having measurable lesion according to RECIST 1.1
5. Life expectancy >3 months
6. Patients must have adequate organ function
7. Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 120 days after last study drug administration. Women of childbearing potential must have a negative pregnancy test ≤ 72 hours prior to Day 1 of study
8. Voluntary informed consent , joining the study with good compliance

Exclusion Criteria:

1. pregnant or lactating women
2. Known history of hypersensitivity to any components of the camrelizumab formulation, or other antibody formulation.
3. Active central nervous system (CNS) metastases with clinical symptoms , including cerebral edema, steroid requirement, or progressive disease.
4. Patients with other malignant tumor within 5 years , except cured skin basal cell carcinoma, cervical carcinoma and Papillary carcinoma of thyroid.
5. Clinically significant cardiovascular diseases
6. Patients have had prior treatment with PD-1/PD-L1 or CTLA-4 antagonists.Received any study drug within 4 weeks prior to the first study drug administration. Enroll in another clinical study, unless it is an observational (non-interventional) clinical study or an intervention follow-up study. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the allergy and nausea, vomiting are allowed. Inhaled or topical use of steroids and adrenocorticosteroid replacement in doses greater than 10mg/ day is permitted in the absence of active autoimmune disease.Patients who have received a live vaccine within 30 days prior to the first study drug administration.Major surgery or major trauma within 4 weeks of first study drug administration. Left ventricular ejection fraction (LVEF) is more than 60% .

(7)Severe infection occurred within 4 weeks before the first first study drug administration (CTC AE > grade 2) (8)Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded. Stable dose of insulin for type 1 diabetes.

(9)History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or organ transplantation and bone marrow transplantation.

(10)Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, pulmonary function damaged seriously etc.

(11)History of active pulmonary tuberculosis infection, or with a history of active pulmonary tuberculosis infection within 1 year prior to enrollment, or with a history of active pulmonary tuberculosis infection prior to 1 year but without formal treatment.

(12)Active hepatitis (transaminase does not meet the inclusion, hepatitis B virus (HBV) DNA ≥10⁴ /ml or hepatitis C virus (HCV) RNA≥103 /ml or higher); Chronic hepatitis B virus carriers who HBV DNA<2000 IU/ml(<104/ml), must receive anti-viral treatment throughout the study.

(13)Known history of psychotropic substance abuse, alcohol abuse and drug abuse.

(14)The investigators did not think the participants were suitable for inclusion.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-03-16 (Estimated); Study Completion 2023-09-16 (Estimated)

PRIMARY OUTCOMES:
tumor cell necrosis rate (TCNR) | 24 months

SECONDARY OUTCOMES:
2 years Overall Survival (OS) rate | 24 months
  The percentage of patients overall survival in 2 years
2 years Progression-free survival (PFS) rate | 24 months
  The percentage of patients Progression-free survival in 2 years
Adverse Events (AEs) | 24 months
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No